CLINICAL TRIAL: NCT04511962
Title: A Feasibility, Randomised Controlled Trial of Tele-rehabilitation Following COVID-19
Brief Title: Feasibility, of Tele-rehabilitation Following COVID-19
Status: Active, not recruiting | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 285205
Record Dates: First submitted 2020-08-05; First posted 2020-08-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Disease
Keywords: rehabilitation, covid19
MeSH Terms: conditions — Lung Diseases; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fast track group: Participants randomised to the fast track group will receive the pulmonary rehabilitation intervention 14 ± 7 days after randomisation.
  Interventions: Other: Tele-Pulmonary rehabilitation
- Wait list group: Participants randomised to the wait-list group will receive the pulmonary rehabilitation intervention 56 ± 7 days after randomisation.
  Interventions: Other: Tele-Pulmonary rehabilitation

INTERVENTIONS:
Other: Tele-Pulmonary rehabilitation — The tele-rehabilitation programme will be delivered via an NHSX / NHS Digital approved commercial video conferencing application. It will comprise an initial assessment followed by 12 bespoke classes delivered by video link over a 6 week period. Participants will be advised to undertake exercises on 5 days each week.

SUMMARY:
Since initial reports of a novel coronavirus emerged from Hubei province, China, the world has been engulfed by a pandemic with over 3 million cases and 225,000 deaths by 30th April 2020. Health care systems around the world have struggled to cope with the number of patients presenting with COVID-19 (the disease caused by the SARS-CoV-2 virus). Although the majority of people infected with the virus have a mild disease, around 20% experience a more severe illness leading to hospital admission and sometimes require treatment in intensive care. People that survive severe COVID-19 are likely to have persistent health problems that would benefit from rehabilitation.

Pulmonary rehabilitation (PR) is a multidisciplinary program which is designed to improve physical and social performance and is typically provided for people with chronic lung conditions. PR courses typically last 6-12 weeks with patients attending classes once or twice weekly and consist of exercise and education components. PR is known to improve symptoms (e.g. breathlessness), quality of life and ability to exercise in those with lung conditions. Breathlessness is a very common symptom reported by people presenting to hospital with COVID-19 and loss of physical fitness will be very common. Using existing pulmonary rehabilitation programmes as a model, we have developed a tele-rehabilitation programme (a programme that will be delivered using video link to overcome the challenges faced by social distancing and shielding advice) for people that have been critically ill with COVID-19. In order to prove whether people benefit from this tele-rehabilitation programme after being admitted to hospital following COVID-19 we would need to perform a large clinical trial. However, before doing this it is important for us to answer some key questions:

* How many people that have been admitted to hospital and needed intensive care treatment for COVID-19 still report breathlessness, fatigue, cough and limitation of activities after being discharged from hospital?
* Is it possible to recruit these people to a trial of tele-rehabilitation after hospital discharge?
* Are people willing and able to perform tele-rehabilitation in their own home using video-link to connect with their therapist?
* Are there other rehabilitation needs that are commonly encountered by people requiring intensive care treatment for COVID-19 that could be addressed by tele-rehabilitation that the programme doesn't currently address? Investigators will perform a small study called a feasibility trial to answer these questions and gather some early information about possible benefits of tele-rehabilitation. Based on our understanding of other similar diseases, doctors and therapists think that people will benefit from rehabilitation after COVID-19. The investigators therefore want to test a trial design that makes sure that everyone gets the treatment. This type of trial is called a feasibility, wait-list design randomised controlled trial. People with breathlessness and some limitation of activities will be selected at random to receive tele-rehabilitation within 2 weeks or to wait 6-8 weeks before starting. how many people were eligible to take part, how many agreed to take part and the symptoms and rehabilitation needs that they have will be assessed. Investigators will then monitor symptoms and ability to exercise at the start and end of the trial and before and after tele-rehabilitation.

DETAILED DESCRIPTION:
STUDY AIMS AND OBJECTIVES Aim: To address the uncertainties relating to the design and conduct of a tele-rehabilitation programme and substantive phase 3 randomised controlled trial to evaluate its effectiveness for people that have been hospitalised with COVID-19 and required additional respiratory support (non-invasive and / or invasive ventilation).

Objectives: Specific study objectives will address uncertainties in four areas.

1. Recruitment: To identify contact:consent ratio, screen failure rate, recruitment and participant retention rate. This will inform the number of sites needed to enrol sufficient participants within an acceptable timeline.
2. Intervention: To assess the acceptability and fidelity of the intervention by measuring adherence in delivery and uptake. Identify additional rehabilitation needs that are not addressed by the tele-rehabilitation programme.
3. Data quality: To assess the amount and pattern of missing data for study measures. Data variability across the range of outcome measures will also be assessed. These findings will inform the choice of primary and secondary outcomes for a definitive trial.
4. Outcome: To assess the best primary outcome and agree other study measures for a definitive trial by identifying i) data completion (objective 3), ii) data variability for potential primary outcome measures to inform sample size calculation for the definitive trial.

In addition to the above feasibility study objectives changes in symptoms, quality of life and measures of functional capacity over time to provide preliminary insights into the natural history of recovery post COVID-19 and potential effect of tele-rehabilitation will be explored.

. STUDY DESIGN Single centre, fast-track (wait-list), randomised controlled feasibility trial of tele-rehabilitation for patients that have been hospitalised with COVID-19 and required non-invasive and/or invasive mechanical ventilation. Patients will be randomised 1:1 to fast-track or wait-list groups using random permuted blocks.

SUMMARY The tele-rehabilitation programme will be delivered by trained therapists and will be structured using conventional pulmonary rehabilitation principles.

Participants will be randomised to fast-track or wait-list groups. All participants will receive the intervention during the course of the trial. Participants randomised to the fast-track group will receive the intervention 14 ± 7 days after randomisation. Participants randomised to the wait-list group will receive the intervention 56 ± 7 days after randomisation.

TELE-REHABILITATION INTERVENTION The tele-rehabilitation programme will be delivered via an NHSX / NHS Digital approved commercial video conferencing application. It will comprise an initial assessment followed by 12 classes delivered by video link over a 6 week period. Participants will be advised to undertake exercises on 5 days each week Participants will be contacted by the interventional physiotherapists prior to commencing the intervention and undertake a virtual (telephone or video) consultation to check eligibility, accessibility and safety to exercise with remote supervision. At this consultation they will be provided with the exercise programme based on their current level of exercise tolerance and functional activity level. Twice a week they will be invited to join a virtual exercise and education group during which the therapists can observe the participants undertaking the exercises. This will allow for safety checks, progression or modifications to be made to the exercises by the therapists. Participants will be taken through a warm up and cool down plus exercise, after which they will be invited to stay to receive educational advice on relevant topics such as managing breathlessness; managing fatigue; diet and hydration; the importance of exercise; returning to the workplace etc. Participants will also be allowed time to share experiences with each other to engender a sense of community and peer support.

ARRANGING THE INTERVENTION Site staff will be trained in local procedures for referral for the intervention. Referral will be undertaken immediately following randomisation and participants informed of their group allocation and start date of the intervention.

Intervention Fidelity Training in the tele-rehabilitation programme will be provided for the therapists involved in intervention delivery. The tele-rehabilitation being delivered has been developed locally as the standard clinical care. For the purpose of the trial, training will be delivered by local therapist familiar with the intervention. A record of staff training in the intervention should be retained in the site file and only those that have received training should be involved in intervention delivery.

Delivery of the intervention should be documented by the delivering therapist within the participant's medical record and CRF. If any components of the intervention are not delivered then the reason for this must be documented in the participant's medical record and CRF.

OUTCOMES AND MEASURES This is a feasibility trial and therefore the primary outcome measures address areas of uncertainty relating to design and delivery of tele-rehabilitation and a Phase 3 randomised controlled trial. These outcomes are termed feasibility outcomes. As part of this trial a number of clinical outcomes will be evaluated with the aim of identifying the most appropriate primary outcome for a subsequent trial and evaluating acceptability and suitability of these measures.

Feasibility Outcomes

The following feasibility outcomes will be assessed:

* Recruitment: Contact to consent ratio; screen failure rate; recruitment rate; retention/follow-up rates at each time point.
* Data quality: completion of clinical outcomes (questionnaires and other assessments) at each time point and patterns of missing data for the study measures.
* Intervention: Adherence in delivery and uptake documented in the clinical record.

Clinical outcomes will be measured and data synthesized to inform the sample size of a definitive trial.

The traffic light system will be used for feasibility outcomes Clinical Outcomes

1. Symptoms

   * The modified Medical research Council Dyspnoea Scale (mMRC) will be used to assess the effect of breathlessness on participants' daily activities. This 5 stage scale measures perceived respiratory disability.
   * Numerical rating scales (NRS, scored 0-10 where 0 = no breathlessness and 10 = worst possible breathlessness) will be used to assess the following aspects of breathlessness over the past 24 hours: best breathlessness / past 24 hours, worst breathlessness / past 24 hours, distress caused by breathlessness / past 24 hours, coping with breathlessness / past 24 hours. The NRS or visual analogue scale (VAS) is recommended as a unidimensional measure of breathlessness in palliative care studies [1]. The NRS is preferable to the 0-100mm VAS [2]. It is highly correlated with VAS scores, but has better test-retest reliability [3, 4], utility [5] and research in pain shows that patients find them easier to use than VAS scales [6]. Although average NRS is often used, we will only use best and worst intensity NRS as "average" has been shown to be prone to "Peak-end" bias [7]. Distress has been used as primary outcomes in trials of breathlessness complex intervention services [8].
   * Cough VAS will be used to assess participants cough.
   * The Modified FACIT-F Scale (version 4) will be used to measure fatigue. This tool has been demonstrated to a valid and reliable tool in a range of malignant and non-malignant diseases including chronic obstructive pulmonary diseae (COPD) [9].
2. Quality of Life The EQ-5D-5L and the EQ visual analogue scale (EQ VAS) will be used to measure participants quality of life. The EQ-5D-5L measures 5 dimensions of health state (mobility, self-care, usual activities, pan/discomfort and anxiety/depression) using 5 levels (no problem, slight problem, moderate problems, severe problems, extreme problems). The EQ VAS asks patients to self-rate their health on a vertical VAS from 'the best health you can imagine' to 'the worst health you can imagine'[10].
3. Mood The hospital anxiety and depression scale (HADS) [11]. The HADS is a short well validated screening assessment tool which will not add unnecessarily to a participant's burden.

   The EQ-5D-5L anxiety and depression domain will also provide insight into participants' mood.
4. Exercise Capacity

The One-Minute Sit-to-Stand Test (STST) assesses the number of times a participant can transition between the sitting and standing positions in a 1 minute period. The STST has shown good correlation with other well validated measures of functional capacity in people with chronic respiratory disease [12] and is suitable for an elderly population [13]. Participants will undertake this assessment in their own homes while observed over a video link. The requirement for specific equipment and space precludes the use of other measures of functional capacity (for example, the 6-minute walk test or incremental shuttle walk test). Other than a chair, the STST requires no specialised equipment and therefore can be undertaken by participants in their own homes.

ELIGIBILITY:
Inclusion Criteria:

1) Males and females aged ≥18 years.

* 2) Suspected or confirmed COVID-19 requiring hospitalisation and either i) non- invasive respiratory support [CPAP, HFNO, NIV] or ii) invasive mechanical ventilation within 3 months of study recruitment.
* 3) > 4 weeks since hospital discharge / first positive COVID-19 swab (whichever is later) at time of screening
* 4) mMRC dyspnoea grades 2 or more.
* 5) Perceived limitation of activities compared with prior to COVID-19 hospitalisation (patient or investigators perception).
* 6) Internet connection and access to a device that supports video calling.
* 7) Able to give informed consent

Exclusion Criteria:

* - 1) Significant comorbid physical or mental illness considered by the investigator to:

  * 2) prevent engagement in modified exercise,
  * 3) impair the participants ability to follow instructions
  * 4) place the participant at undue risk during exercise training
  * 5) adversely affect the recovery or rehabilitation trajectory
* Unwilling or unable to consent or complete study measures.
* Current involvement in other interventional clinical trials relating to COVID-19 (e.g. clinical trial of an investigational medicinal product)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified from those patients being contacted post hospitalisation at Hull University Teaching Hospitals NHS Trust due to Covid-19. Patients selected will be those still reporting breathlessness, fatigue, cough and limited activity.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment - contact to consent ratio | through study completion an average of a year
  The proportion of the total patients contacted, that meet the intieligibility criteria and give consent to take part
  * Data quality: completion of clinical outcomes (questionnaires and other assessments) at each time point and patterns of missing data for the study measures.
  * Intervention: Adherence in delivery and uptake documented in the clinical record.
Recruitment - screen failure rate | through study completion an average of a year
  The proportion of patients consented to the study that do not meet the eligibility criteria
Recruitment rate | through study completion an average of a year
  The number patients recruited over the designated time frame
Recruitment retention | through study completion an average of 16 months
  The proportion of consented patients that complete the study

SECONDARY OUTCOMES:
The Modified Medical Research Council (MMRC) Dyspnoea Scale | 8 weeks
  The Modified Medical Research Council Dyspnoea Scale is a self rating tool to measure the degree of disability that breathlessness poses on day to day activities on a scale of 0-4; the higher the score the worse the outcome. A comparison of Change in MMRC dyspnoea scale from baseline to post 8 weeks tele rehab within the group and between fast track and wait list group.
Numerical Rating Scale (NRS) of breathlessness | 8 weeks
  The Numerical Rating Scale is a self rating tool to measure breathlessness on a 0-10 scale; a higher number indicates a worse outcome. A comparison of change in numerical scale from baseline to post 8 weeks tele rehab within the group and between fast track and wait list group
Cough Visual analogue Scale (VAS) | 8 weeks
  The Cough Visual Analogue Scale is a self rating assessment of cough on an 0-100mm scale: the higher the number reported the worse the symptom. A comparison of Change in cough visual analogue scale from baseline to post 8 weeks tele rehab within the group and between fast track and wait list group
EQ-5D-5L questionnaire | 8 weeks
  The EQ-5D-5L questionnaire assesses the patients current health status and consists of two elements: 1. Visual Analogue Scale with a range of 0-100mm- the higher the number the worse the outcome 2. A quality of life questionnaire split into 5 domains which generates a 5 digit code ranging from 11111 to 55555 with the higher number indicating a worse outcome. A comparison of Change in EQ-5D-5L quality of life questionnaire from baseline to post 8 weeks tele rehab within the group and between fast track and wait list group
Hospital Anxiety and Depression scale | 8 weeks
  The Hospital Anxiety and Depression scale consists of two sub scales anxiety and depression with a range of between 0-21, the higher score indicating the worse outcome. A comparison of Change in Hospital anxiety and depression questionnaire from baseline to post 8 weeks tele rehab within the group and between fast track and wait list group
Sit to stand test | 8 weeks
  comparison of sit to stand test from baseline to post 8 weeks tele rehab within the group and between fast track and wait list grou

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital, Cottingham, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dorman S, Jolley C, Abernethy A, Currow D, Johnson M, Farquhar M, Griffiths G, Peel T, Moosavi S, Byrne A, Wilcock A, Alloway L, Bausewein C, Higginson I, Booth S. Researching breathlessness in palliative care: consensus statement of the National Cancer Research Institute Palliative Care Breathlessness Subgroup. Palliat Med. 2009 Apr;23(3):213-27. doi: 10.1177/0269216309102520. Epub 2009 Feb 27. PMID 19251835
- [Background] Powers J, Bennett SJ. Measurement of dyspnea in patients treated with mechanical ventilation. Am J Crit Care. 1999 Jul;8(4):254-61. PMID 10392226
- [Background] Wilcock A, Crosby V, Clarke D, Tattersfield A. Repeatability of breathlessness measurements in cancer patients. Thorax. 1999 Apr;54(4):375. doi: 10.1136/thx.54.4.374b. No abstract available. PMID 10400541
- [Background] Gift AG, Narsavage G. Validity of the numeric rating scale as a measure of dyspnea. Am J Crit Care. 1998 May;7(3):200-4. PMID 9579246
- [Background] Booth S, Galbraith S, Ryan R, Parker RA, Johnson M. The importance of the feasibility study: Lessons from a study of the hand-held fan used to relieve dyspnea in people who are breathless at rest. Palliat Med. 2016 May;30(5):504-9. doi: 10.1177/0269216315607180. Epub 2015 Oct 22. PMID 26494368
- [Background] Caraceni A. Evaluation and assessment of cancer pain and cancer pain treatment. Acta Anaesthesiol Scand. 2001 Oct;45(9):1067-75. doi: 10.1034/j.1399-6576.2001.450903.x. PMID 11683654
- [Background] Wade J, Mendonca S, Booth S, Ewing G, Gardener AC, Farquhar M. Are within-person Numerical Rating Scale (NRS) ratings of breathlessness 'on average' valid in advanced disease for patients and for patients' informal carers? BMJ Open Respir Res. 2017 Oct 11;4(1):e000235. doi: 10.1136/bmjresp-2017-000235. eCollection 2017. PMID 29071084
- [Background] Farquhar MC, Prevost AT, McCrone P, Brafman-Price B, Bentley A, Higginson IJ, Todd C, Booth S. Is a specialist breathlessness service more effective and cost-effective for patients with advanced cancer and their carers than standard care? Findings of a mixed-method randomised controlled trial. BMC Med. 2014 Oct 31;12:194. doi: 10.1186/s12916-014-0194-2. PMID 25358424
- [Background] Al-shair K, Muellerova H, Yorke J, Rennard SI, Wouters EF, Hanania NA, Sharafkhaneh A, Vestbo J; ECLIPSE investigators. Examining fatigue in COPD: development, validity and reliability of a modified version of FACIT-F scale. Health Qual Life Outcomes. 2012 Aug 23;10:100. doi: 10.1186/1477-7525-10-100. PMID 22913289
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Ozalevli S, Ozden A, Itil O, Akkoclu A. Comparison of the Sit-to-Stand Test with 6 min walk test in patients with chronic obstructive pulmonary disease. Respir Med. 2007 Feb;101(2):286-93. doi: 10.1016/j.rmed.2006.05.007. Epub 2006 Jun 27. PMID 16806873
- [Background] Gross MM, Stevenson PJ, Charette SL, Pyka G, Marcus R. Effect of muscle strength and movement speed on the biomechanics of rising from a chair in healthy elderly and young women. Gait Posture. 1998 Dec 1;8(3):175-185. doi: 10.1016/s0966-6362(98)00033-2. PMID 10200407